CLINICAL TRIAL: NCT01092286
Title: Effect of Neuromuscular Warm-up on Injuries in Female Athletes in Urban Public High Schools: A Cluster-randomized Controlled Trial
Brief Title: Effect of Neuromuscular Warm-up on Injuries in Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Cynthia LaBella, Medical Director, Institute for Sports Medicine, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB2006-12888
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Knee Injuries; Anterior Cruciate Ligament Injuries; Ankle Injuries; Lower Extremity Injuries
Keywords: Knee injury; ankle sprain; anterior cruciate ligament; adolescent; soccer; basketball; prevention
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries; Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- neuromuscular warm-up (Experimental): coaches in this arm use the prescribed warm-up before team practices
  Interventions: Other: neuromuscular warm-up
- no warm-up (No Intervention): coaches use their usual warm-up before team practices

INTERVENTIONS:
Other: neuromuscular warm-up — neuromuscular warm-up exercises that take 20 minutes to perform
  Other Names: Knee Injury Prevention Program (KIPP)
  Arms: neuromuscular warm-up

SUMMARY:
The goal of the study is to determine effect of coach-led neuromuscular warm-up on non-contact, lower extremity (LE) injury rates among female athletes in a predominantly non-white public high school system. The investigators hypothesized the warm-up would reduce non-contact LE injuries.

DETAILED DESCRIPTION:
We will recruit basketball and soccer coaches and their athletes from Chicago public high schools. We will randomize teams to intervention and control groups. We will train intervention coaches to implement a 20-minute neuromuscular warm-up and tracked training costs. Control coaches will use their usual warm-up. All coaches will report weekly athlete exposures (AEs) and injuries resulting in a missed practice/game. Research assistants will interview injured athletes. We will compare injury rates between control and intervention groups.

ELIGIBILITY:
Inclusion Criteria for High School Students (initial part of study - completed)

* plays basketball or soccer for a Chicago public high school team
* coaches basketball or soccer for a Chicago public high school team
* female, age 14-20

Inclusion Criteria for coaches (current part of study):

* Willing to implement a new warm-up before their team's practices and games
* Willing to complete a pre- and post-season survey before and after using the warm-up program for one season (surveys are attached).
* Willing to complete a pre- and post-workshop test before and after the workshop (tests are attached).
* Willing to allow study personnel to observe their implementation of the warm-up at up to three team practices or games.

Exclusion Criteria for coaches (current part of study) There are no separate exclusion criteria for coaches.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1653 (Actual)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
lower extremity injury rates | one year

SECONDARY OUTCOMES:
coach compliance with warm-up | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R LaBella, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] LaBella CR, Huxford MR, Grissom J, Kim KY, Peng J, Christoffel KK. Effect of neuromuscular warm-up on injuries in female soccer and basketball athletes in urban public high schools: cluster randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Nov;165(11):1033-40. doi: 10.1001/archpediatrics.2011.168. PMID 22065184